CLINICAL TRIAL: NCT04328558
Title: The Effectiveness of Clavipectoral Fascia Plane Block for Analgesia After Clavicle Surgery: Randomized, Prospective Study
Brief Title: Clavipectoral Fascia Plane Block for Clavicle Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 10
Record Dates: First submitted 2020-03-28; First posted 2020-03-31 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Clavicle Injury; Clavicle Fracture
Keywords: Clavicle fracture; Clavipectoral fascia plane block; Postoperative analgesia

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is clavipectoral fascia plane block group. The second one is no intervention control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CPB = Clavipectoral fascia plane block group (Active Comparator): In group CPB, CPB will be performed with patients in the supine position. The probe will be placed on the anterior border of the medial third of the clavicle. A 22-gauge block needle will be inserted in a caudal to cephalic direction, the periosteum of the clavicle and the surrounding fascia will be visualized, 20 ml of 0.25% bupivacaine will be injected between these two layers. The local anesthetic spread to medial and lateral third of the clavicle will be seen.
  Interventions: Other: Clavipectoral fascia plane block group
- Group C = Control group (No Intervention): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.

INTERVENTIONS:
Other: Clavipectoral fascia plane block group — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.
  Arms: Group CPB = Clavipectoral fascia plane block group

SUMMARY:
The pain after clavicle fracture surgery may be managed with combined superficial cervical plexus-interscalene block and recently clavipectoral fascia plane block (CPB). CPB was defined by Valdes in 2017 firstly. It may be used for postoperative analgesia after clavicle surgery. CPB may be an alternative to interscalene brachial plexus block.

The aim of this study is to evaluate the efficacy of the US-guided CPB for postoperative analgesia management compare to no intervention control group after clavicle surgery. The primary aim is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting).

DETAILED DESCRIPTION:
Clavicle fracture is common in men and children after a direct fall on shoulder during sport activity such as cycling or an injury during a traffic accident. The pain after clavicle fracture surgery may be managed with combined superficial cervical plexus-interscalene block and recently clavipectoral fascia plane block (CPB). CPB was defined by Valdes in 2017 firstly. It may be used for postoperative analgesia after clavicle surgery. The clavipectoral fascia covers the clavicular site of the pectoralis major muscle. It provides the potential interfascial space between the clavicle and the pectoralis major muscle. CPB provide effective analgesia after clavicle surgery. It is also easy to perform. With this advantage and its analgesic effectiveness for clavicle surgery, CPB may be an alternative to interscalene brachial plexus block. However, randomized clinical efficacy trials are needed to investigate the effectiveness of CPB for clavicle fractures. In the literature, data about CPB is so limited, however it seems a good alternative to brachial plexus block for pain management after clavicle fracture The aim of this study is to evaluate the efficacy of the US-guided CPB for postoperative analgesia management compare to no intervention control group after clavicle surgery. The primary aim is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for clavicle surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | Change from baseline opioid consumption at postoperative 1, 2, 4, 8, 16, 24 and 48 hours
  The primary aim is to compare postoperative opioid consumption

SECONDARY OUTCOMES:
Pain scores (Visual analogue scores-VAS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16, and 24 hours.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Atalay YO, Mursel E, Ciftci B, Iptec G. Clavipectoral Fascia Plane Block for Analgesia after Clavicle Surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2019 Dec;66(10):562-563. doi: 10.1016/j.redar.2019.06.006. Epub 2019 Nov 11. No abstract available. English, Spanish. PMID 31727320
- [Background] Ince I, Kilicaslan A, Roques V, Elsharkawy H, Valdes L. Ultrasound-guided clavipectoral fascial plane block in a patient undergoing clavicular surgery. J Clin Anesth. 2019 Dec;58:125-127. doi: 10.1016/j.jclinane.2019.07.011. Epub 2019 Aug 1. No abstract available. PMID 31377668
- [Background] Ueshima H, Ishihara T, Hosokawa M, Otake H. RETRACTED: Clavipectoral fascial plane block in a patient with dual antiplatelet therapy undergoing emergent clavicular surgery. J Clin Anesth. 2020 May;61:109648. doi: 10.1016/j.jclinane.2019.109648. Epub 2019 Nov 13. No abstract available. PMID 31732427 (Retraction: PMID 35393209 J Clin Anesth. 2022 Aug;79:110779)